CLINICAL TRIAL: NCT01315132
Title: A Two Step Approach To Matched-Sibling Allogeneic Hematopoietic Stem Cell Transplantation for High-Risk Hematological Malignancies
Brief Title: A Study of Bone Marrow Transplantation Using Fully-Matched Relatives as Donors for Patients With Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08D.85; 2007-61 (Other: CCRRC); JT 1275 (Other: JeffTrial Number)
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hematological Malignancies; Leukemia; Lymphoma; Multiple Myeloma; Hodgkin's Disease
Keywords: Myeloablative Hematopoietic Stem Cell Transplant; Cyclophosphamide tolerization; 2 Step Approach; Hematological malignancies; leukemia; lymphoma; multiple myeloma; Hodgkin's Disease
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Transplantation (Experimental): Matched Sibling Allogeneic Transplantation
  Interventions: Device: Matched Sibling Allogeneic Transplantation

INTERVENTIONS:
Device: Matched Sibling Allogeneic Transplantation — Patients undergoing myeloablative hematopoietic stem cell transplant from HLA identical related donors using cyclophosphamide tolerization
  Other Names: CliniMACS

SUMMARY:
This research study uses a drug called cyclophosphamide to decrease the incidence of GVHD in matched sibling hematopoietic stem cell transplant. In doing so, the goal of the study is to increase overall survival.

DETAILED DESCRIPTION:
This research protocol has been developed for patients undergoing matched-sibling hematopoietic stem cell transplant (HSCT). The patients who are treated according to this 2 step allogeneic HSCT protocol will receive cyclophosphamide to induce in-vivo tolerization of both autologous and allogeneic lymphocytes, followed by an allogeneic CD34-selected HSCT. The primary research questions relate to immune reconstitution, incidence of GVHD, and relapse in patients who receive lymphocyte treatment of this type in allogeneic HSCT and how it impacts overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a hematologic or oncologic diagnosis in which allogeneic HSCT is thought to be beneficial, and in whom front-line therapy has already been applied. Patients will be considered high-risk if they have any of the following:

   1. Age > 50 years
   2. ECOG Performance status of <2
   3. Acute leukemia: requiring more than one chemotherapy regimen to obtain 1st CR; second or greater CR, 1st relapse; any ph+ ALL
   4. CML 2nd chronic phase, accelerated phase, or blastic phase
   5. MDS with IPS of Intermediate 2 or greater
   6. Any myeloproliferative disorder
   7. Hodgkin lymphoma: relapsed, refractory, or primary induction failure
   8. Non-Hodgkin lymphoma: relapsed, refractory, primary treatment failure, or not eligible for an autologous HSCT
   9. Other conditions not listed will be assessed as high-risk by the PI
2. Patients must have a related donor who is either HLA-identical or a one antigen mismatch at the HLA- A; B; C; and DR loci.
3. Patients must adequate organ function:

   1. LVEF of >45%
   2. DLCO (adjusted for hemoglobin) >45% of predicted
   3. Adequate liver function as defined by a serum bilirubin <1.8, AST or ALT < 2.5X upper limit of normal
   4. Creatinine clearance of > 60 ml/min
4. Patients must be willing to use contraception if they have childbearing potential
5. Able to give informed consent

Exclusion Criteria:

1. ECOG performance status of 3 or 4.
2. HIV positive
3. Active involvement of the central nervous system with malignancy
4. Psychiatric disorder that would preclude patients from signing an informed consent
5. Pregnancy
6. Patients with life expectancy of < 6 months for reasons other than their underlying hematologic/oncologic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-04-10 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Flomenberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allogeneic Transplantation
Started | 47
Completed | 46
Not Completed | 1
Not completed — not treated due to disease progression | 1

BASELINE CHARACTERISTICS:
Population: While 47 participants were enrolled, one participant was removed from the study prior to treatment and will not be counted in the outcomes of the trial
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 37
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Overall Survival
Description: The primary objective of this prospective, phase II trial was to obtain an OS rate of >60% at 1 year in patients undergoing a 2 step HSCT from an HLA compatible family donor. The >60% threshold was selected as a composite efficacy measure as patients with any hematologic diagnosis, stage of disease, or age as old as 65 years were eligible for this treatment protocol.
Time Frame: 1 Year after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 46
Participants | 41

2. Secondary Outcome: Graft Versus Host Disease (GVHD)
Time Frame: 1 Year after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Transplantation
Number analyzed (Participants) | 46
Participants
  Acute GVHD | 6
  Chronic GVHD | 4
  No GVHD | 36

ADVERSE EVENTS:
Time Frame: from baseline through one year after transplant
Arm/Group | Allogeneic Transplantation
All-Cause Mortality (participants affected / at risk) | 16/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 32/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Transplantation (N=46)
Mucositis (Gastrointestinal disorders) | 32 (32)
Diarrhea (Gastrointestinal disorders) | 30 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT01315132/Prot_SAP_000.pdf